CLINICAL TRIAL: NCT00634933
Title: A Randomized, Parallel, Double-Blind, Placebo-Controlled Dose Regimen Finding Study To Evaluate The Safety And Efficacy Of TRU-015 In Subjects With Active Seropositive Rheumatoid Arthritis On A Stable Background Of Methotrexate
Brief Title: Study Evaluating 2 Dosing Regimens Of TRU-015 In Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on 21 June 2010 due to results not meeting the primary endpoint. No safety reasons contributed to the termination of the study.
Sponsor: Pfizer (Industry)
Collaborators: Trubion Pharmaceuticals/Emergent BioSolutions Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3206K1-2203; B2051001; NCT01616706 (obsolete NCT alias)
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-02

CONDITIONS: Arthritis, Rheumatoid
Keywords: active; rheumatoid; arthritis; anti CD20
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity; Arthritis | interventions — TRU-015 protein; Methylprednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Consists of Arms 1a and 1b
  Interventions: Drug: TRU-015; Drug: Methylprednisolone; Drug: Prednisone
- Arm 2 (Experimental): Consists of Arms 2a and 2b
  Interventions: Drug: TRU-015; Drug: Methylprednisolone; Drug: Prednisone
- Arm 3 (Placebo Comparator): Consists of Arms 3a and 3b.
  Interventions: Drug: TRU-015; Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: TRU-015 — IV 800 mg TRU-015 at Baseline (both arms) and Week 24 (both arms); corresponding IV Placebo at Week 12 and Week 36 (both arms).
  Arms: Arm 1
Drug: Methylprednisolone — IV 100 mg Methylprednisolone at Baseline (both arms), Week 12 (arm 1a) and Week 24 (both arms); corresponding IV Placebo at Week 12 (Arm 1b) and Week 36 (both arms).
  Arms: Arm 1
Drug: Prednisone — Oral 20 mg tablets Prednisone at Baseline (both arms), Week 12 (arm 1a), and Week 24 (both arms); corresponding Oral Placebo at Week 12 (Arm 1b) and Week 36 (both arms)
  Arms: Arm 1
Drug: TRU-015 — IV 800 mg TRU-015 at Baseline (both arms), Week 12 (both arms), and Week 36 (both arms); corresponding IV Placebo at Week 24 (both arms).
  Arms: Arm 2
Drug: Methylprednisolone — IV 100 mg Methylprednisolone at Baseline (both arms), Week 12 (both arms), and Week 36 (both arms); corresponding IV Placebo at Week 36 (both arms).
  Arms: Arm 2
Drug: Prednisone — Oral 20 mg tablets Prednisone at Baseline (both arms), Week 12 (arm 2a) and Week 36 (both arms); corresponding Oral Placebo at Week 12 (Arm 2b) and Week 24 (both arms).
  Arms: Arm 2
Drug: TRU-015 — IV 800 mg TRU-015 at Week 24 (both arms) and Week 36 (arm 3a); corresponding IV Placebo at Baseline (both arms), Week 12 (both arms) and Week 36 (arm 3b).
  Arms: Arm 3
Drug: Methylprednisolone — IV 100 mg Methylprednisolone at Baseline (both arms), Week 12 (arm 3a), Week 24 (both arms), and Week 36 (arm 3a); corresponding IV Placebo at Week 12 (arm 3b) and Week 36 (arm 3b).
  Arms: Arm 3
Drug: Prednisone — Oral 20 mg tablets Prednisone at Baseline (both arms), Week 12 (arm 3a), Week 24 (both arms) and Week 36 (arm 3a); corresponding Oral Placebo at Week 12 (Arm 3b) and Week 36 (arm 3b).
  Arms: Arm 3

SUMMARY:
This study will evaluate the efficacy and safety of two dosing regimens of a compound known as TRU-015 in combination with methotrexate (MTX) in patients with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of active seropositive rheumatoid arthritis on a stable dose of methotrexate (7.5-25 mg weekly) for at least 12 weeks with or without a history of anti-TNF use.

Exclusion Criteria:

* Any prior use of rituximab or other B cell depleting agents.
* Any significant health problem other than rheumatoid arthritis
* Clinically significant laboratory abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (27):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Paradise Valley, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Maria, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Grande Rapids, Michigan
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Mayfield Village, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Danville, Pennsylvania
  - Pfizer Investigational Site, State College, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Wilkes-Barre, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Clarksburg, West Virginia
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Liège
- Canada (6):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Sydney, Nova Scotia
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Trois-Rivières, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- France (3):
  - Pfizer Investigational Site, Montpellier, France
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Toulouse
- Germany (4):
  - Pfizer Investigational Site, Vogelsang, Gommern
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Würzburg
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Nyíregyháza
- Mexico (5):
  - Pfizer Investigational Site, Mexicali, Baja California/Mexico
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Morelia, Michoacán
  - Pfizer Investigational Site, Culiacán, Sinaloa/Mexico
  - Pfizer Investigational Site, Mexico City
- Pfizer Investigational Site, Leiden, Netherlands
- Romania (4):
  - Pfizer Investigational Site, Iași, Iaşi
  - Pfizer Investigational Site, Bucharest, Romania
  - Pfizer Investigational Site, Cluj-Napoca, Romania
  - Pfizer Investigational Site, Bucharest
- Serbia (2):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Niška Banja

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3206K1-2203&StudyName=Study%20Evaluating%202%20Dosing%20Regimens%20Of%20TRU-015%20In%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo infusion, matched to TRU-015 (800 milligram [mg]), intravenously (IV) along with methylprednisolone 100 mg IV 1 hour (hr) prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at baseline. Placebo infusion, matched to TRU-015 (800 mg), IV along with methylprednisolone 100 mg or matching placebo IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of the infusion at Week 12. Participants in this group were assigned to either Placebo/TRU-SD or Placebo/TRU-ID in the Part B of the study.
- TRU-015 Single Dose: TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at baseline. Placebo infusion, matched to TRU-015 800 mg, IV, methylprednisolone 100 mg or matching placebo IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of infusion at Week 12. TRU-015 800 mg infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 24. Placebo infusion, matched to TRU-015 (800 mg) IV along with placebo matched to methylprednisolone 100 mg IV 1 hr prior to infusion and placebo matched to prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 36.
- TRU-015 Induction Dose: TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at baseline. TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of infusion at Week 12. Placebo infusion, matched to TRU-015 (800 mg), IV, placebo matched to methylprednisolone 100 mg IV 1 hr prior to infusion and placebo capsule matched to prednisone 20 mg orally each day for 2 days prior to and on the morning of infusion at Week 24. TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 36.
- Placebo/TRU-015 Single Dose: TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 24. Placebo infusion, matched to TRU-015 (800 mg), IV, placebo matched to methylprednisolone 100 mg IV 1 hr prior to infusion and placebo capsule matched to prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 36.
- Placebo/TRU-015 Induction Dose: TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 24 and 36.
Period: Part A: Baseline to Week 24
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose | Placebo/TRU-015 Single Dose | Placebo/TRU-015 Induction Dose
Started | 74 | 75 | 73 | 0 | 0
Completed | 63 | 57 | 55 | 0 | 0
Not Completed | 11 | 18 | 18 | 0 | 0
Not completed — Adverse Event | 4 | 4 | 8 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Failed to Return | 1 | 0 | 0 | 0 | 0
Not completed — Investigator Request | 1 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 3 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 8 | 5 | 0 | 0
Period: Between Part A and Part B
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose | Placebo/TRU-015 Single Dose | Placebo/TRU-015 Induction Dose
Started | 0 | 57 | 55 | 31 | 32
Completed | 0 | 56 | 55 | 31 | 32
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Period: Part B: Week 24 to Week 52
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose | Placebo/TRU-015 Single Dose | Placebo/TRU-015 Induction Dose
Started | 0 | 56 | 55 | 31 | 32
Completed | 0 | 42 | 33 | 25 | 22
Not Completed | 0 | 14 | 22 | 6 | 10
Not completed — Adverse Event | 0 | 1 | 1 | 1 | 0
Not completed — Discontinuation of Study by Sponsor | 0 | 11 | 14 | 3 | 7
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo infusion, matched to TRU-015 (800 mg), IV along with methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at baseline. Placebo infusion, matched to TRU-015 (800 mg), IV along with methylprednisolone 100 mg or matching placebo IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of the infusion at Week 12. TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 24. TRU-015 (800 mg) infusion or matching placebo IV, methylprednisolone 100 mg or matching placebo IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of infusion at Week 36.
- TRU-015 Single Dose: TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at baseline. Placebo infusion, matched to TRU-015 (800 mg), IV, methylprednisolone 100 mg or matching placebo IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of infusion at Week 12. TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 24. Placebo infusion, matched to TRU-015 (800 mg) IV along with placebo matched to methylprednisolone 100 mg IV 1 hr prior to infusion and placebo matched to prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 36.
- Total: Total of all reporting groups
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose | Total
Number analyzed (Participants) | 74 | 75 | 73 | 222
Age Continuous [Mean (Standard Deviation); unit: years] | 50.62 (11.07) | 52.99 (11.33) | 52.55 (13.00) | 52.05 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 62 | 59 | 185
  Male | 10 | 13 | 14 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR 50) Response at Week 24
Description: ACR50 response: greater than or equal to (>=) 50 percent (%) improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ-DI]); and C-Reactive Protein (CRP).
Time Frame: Week 24
Population: Modified intent-to-treat (mITT) population included all randomized participants who received any portion of test article. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
percentage of participants | 16.2 | 29.3 | 27.4
Statistical Analysis 1: Comparison: Placebo vs TRU-015 Single Dose; A 2-sided Cochran-Mantel-Haenszel test (CMH), stratified by prior anti-tumor necrosis factor (anti-TNF) use and geographic region, was used; Test type: Superiority or Other; p = 0.061, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs TRU-015 Induction Dose; A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.120, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: >= 20% improvement in tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (HAQ-DI); and CRP.
Time Frame: Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: mITT population included all randomized participants who received any portion of test article. LOCF method was used to impute missing values. Data for time points after Week 24 were not analyzed because of early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
percentage of participants
  Week 2 | 17.6 | 21.3 | 26.0
  Week 4 | 31.1 | 34.7 | 34.2
  Week 8 | 31.1 | 44.0 | 42.5
  Week 12 | 31.1 | 52.0 | 49.3
  Week 16 | 41.9 | 64.0 | 61.6
  Week 20 | 47.3 | 62.7 | 64.4
  Week 24 | 43.2 | 61.3 | 67.1
Statistical Analysis 1: Comparison: Placebo vs TRU-015 Single Dose; Week 2: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.570, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs TRU-015 Induction Dose; Week 2: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.200, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs TRU-015 Single Dose; Week 4: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.616, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs TRU-015 Induction Dose; Week 4: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.671, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs TRU-015 Single Dose; Week 8: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.108, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs TRU-015 Induction Dose; Week 8: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.174, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs TRU-015 Single Dose; Week 12: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs TRU-015 Induction Dose; Week 12: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.029, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs TRU-015 Single Dose; Week 16: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Placebo vs TRU-015 Induction Dose; Week 16: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Placebo vs TRU-015 Single Dose; Week 20: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.062, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Placebo vs TRU-015 Induction Dose; Week 20: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.049, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Placebo vs TRU-015 Single Dose; Week 24: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.030, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Placebo vs TRU-015 Induction Dose; Week 24: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: >=50% improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (HAQ-DI); and CRP.
Time Frame: Week 2, 4, 8, 12, 16, 20, 28, 32, 36, 40, 44, 48, 52
Population: mITT population included all randomized participants who received any portion of test article. LOCF method was used to impute missing values. Data for time points after Week 20 were not analyzed because of early termination of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
percentage of participants
  Week 2 | 0.0 | 8.0 | 6.8
  Week 4 | 6.8 | 8.0 | 6.8
  Week 8 | 12.2 | 10.7 | 8.2
  Week 12 | 14.9 | 16.0 | 13.7
  Week 16 | 16.2 | 30.7 | 31.5
  Week 20 | 16.2 | 28.0 | 28.8
Statistical Analysis 1: Comparison: Placebo vs TRU-015 Single Dose; Week 2: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs TRU-015 Induction Dose; Week 2: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs TRU-015 Single Dose; Week 4: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.794, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs TRU-015 Induction Dose; Week 4: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.966, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs TRU-015 Single Dose; Week 8: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.770, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs TRU-015 Induction Dose; Week 8: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.456, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs TRU-015 Single Dose; Week 12: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.880, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs TRU-015 Induction Dose; Week 12: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.814, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs TRU-015 Single Dose; Week 16: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.042, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Placebo vs TRU-015 Induction Dose; Week 16: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Placebo vs TRU-015 Single Dose; Week 20: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.086, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Placebo vs TRU-015 Induction Dose; Week 20: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.082, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (HAQ-DI); and CRP.
Time Frame: Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
percentage of participants
  Week 2 | 0.0 | 1.3 | 1.4
  Week 4 | 1.4 | 1.3 | 0.0
  Week 8 | 1.4 | 2.7 | 1.4
  Week 12 | 1.4 | 2.7 | 2.7
  Week 16 | 6.8 | 8.0 | 6.8
  Week 20 | 2.7 | 6.7 | 6.8
  Week 24 | 2.7 | 9.3 | 9.6
Statistical Analysis 1: Comparison: Placebo vs TRU-015 Single Dose; Week 2: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.325, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs TRU-015 Induction Dose; Week 2: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.338, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs TRU-015 Single Dose; Week 4: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.983, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs TRU-015 Induction Dose; Week 4: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.296, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs TRU-015 Single Dose; Week 8: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.575, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs TRU-015 Induction Dose; Week 8: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs TRU-015 Single Dose; Week 12: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.573, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs TRU-015 Induction Dose; Week 12: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.563, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs TRU-015 Single Dose; Week 16: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.768, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Placebo vs TRU-015 Induction Dose; Week 16: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.977, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Placebo vs TRU-015 Single Dose; Week 20: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.249, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Placebo vs TRU-015 Induction Dose; Week 20: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.268, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Placebo vs TRU-015 Single Dose; Week 24: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.089, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Placebo vs TRU-015 Induction Dose; Week 24: A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.079, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Tender Joints
Description: The number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
tender joints
  Baseline | 17.0 (6.1) | 16.8 (7.0) | 17.7 (6.2)
  Week 2 | 13.6 (7.0) | 11.9 (7.4) | 13.0 (7.7)
  Week 4 | 11.9 (7.0) | 10.7 (7.7) | 11.6 (7.7)
  Week 8 | 11.7 (8.4) | 9.8 (6.7) | 10.1 (7.4)
  Week 12 | 11.0 (7.9) | 8.8 (6.9) | 9.6 (7.7)
  Week 16 | 9.4 (7.9) | 7.3 (7.0) | 8.4 (7.2)
  Week 20 | 9.0 (7.2) | 7.6 (7.3) | 7.6 (7.1)
  Week 24 | 9.4 (7.5) | 8.1 (7.6) | 7.6 (7.4)

6. Secondary Outcome: Number of Swollen Joints
Description: The number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: Baseline. Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
swollen joints
  Baseline | 12.2 (4.4) | 12.3 (6.0) | 13.9 (5.7)
  Week 2 | 9.5 (5.7) | 9.0 (6.5) | 10.2 (6.2)
  Week 4 | 7.8 (5.3) | 8.5 (6.4) | 9.0 (6.2)
  Week 8 | 7.0 (5.7) | 6.9 (5.2) | 7.7 (5.6)
  Week 12 | 7.6 (5.8) | 6.0 (4.9) | 7.1 (5.5)
  Week 16 | 6.1 (5.4) | 5.1 (5.2) | 5.9 (4.7)
  Week 20 | 6.0 (5.4) | 4.8 (4.6) | 5.1 (4.9)
  Week 24 | 6.2 (5.5) | 4.7 (4.6) | 5.0 (5.0)

7. Secondary Outcome: Duration of Morning Stiffness
Description: Duration of morning stiffness is defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (if none was present = 0; if morning stiffness was continuing, average of duration of stiffness over the past 3 days was reported; if stiffness persisted the entire day, 1440 minutes [24 hours*60 minutes] was recorded).
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Data was not analyzed because development of TRU-015 was discontinued as results of primary analysis did not meet the predefined efficacy criteria.
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Visual Analogue Scale for Pain (VAS-pain)
Description: 100 millimeter (mm) line (Visual Analog Scale) marked by participant. Intensity of pain range (over past week): 0 = no pain to 100 = worst possible pain.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
mm
  Baseline | 65.4 (17.9) | 62.5 (20.7) | 61.6 (23.0)
  Week 2 | 53.0 (21.2) | 47.7 (25.2) | 49.6 (24.6)
  Week 4 | 53.6 (20.3) | 48.9 (25.9) | 49.0 (24.2)
  Week 8 | 56.4 (23.0) | 45.8 (24.0) | 47.0 (24.5)
  Week 12 | 54.3 (21.6) | 42.3 (24.1) | 44.8 (25.4)
  Week 16 | 51.1 (24.2) | 39.3 (24.4) | 40.8 (25.2)
  Week 20 | 51.1 (21.6) | 39.5 (24.2) | 39.1 (25.7)
  Week 24 | 49.2 (22.2) | 39.2 (25.0) | 43.9 (28.3)

9. Secondary Outcome: Physician Global Assessment (PGA) of Disease Activity
Description: Physician Global Assessment of Disease Activity was measured on a 0 to 10 point scale, where 0 = no disease activity and 10 = extreme disease activity.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
units on a scale
  Baseline | 6.8 (1.3) | 6.4 (1.6) | 6.6 (1.7)
  Week 2 | 5.5 (1.5) | 5.1 (2.2) | 5.2 (1.9)
  Week 4 | 5.0 (1.9) | 5.0 (2.3) | 4.9 (2.1)
  Week 8 | 5.0 (2.2) | 4.1 (2.1) | 4.4 (2.1)
  Week 12 | 4.8 (2.1) | 4.1 (2.1) | 4.3 (2.3)
  Week 16 | 4.6 (2.4) | 3.7 (2.1) | 3.6 (2.1)
  Week 20 | 4.4 (2.1) | 3.8 (1.8) | 3.6 (2.2)
  Week 24 | 4.3 (2.2) | 3.7 (2.1) | 3.6 (2.4)

10. Secondary Outcome: Patient Global Assessment (PtGA) of Disease Activity
Description: Measured using a 0-10 point scale, where 0 = no disease activity and 10 = extreme disease activity.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
units on a scale
  Baseline | 7.3 (1.6) | 6.9 (1.9) | 7.0 (2.3)
  Week 2 | 6.2 (2.1) | 5.6 (2.4) | 5.6 (2.3)
  Week 4 | 6.0 (1.8) | 5.4 (2.4) | 5.6 (2.4)
  Week 8 | 6.2 (2.1) | 5.2 (2.4) | 5.3 (2.3)
  Week 12 | 5.9 (2.1) | 4.8 (2.3) | 5.2 (2.4)
  Week 16 | 6.6 (9.2) | 4.4 (2.3) | 4.6 (2.5)
  Week 20 | 5.5 (2.1) | 4.5 (2.3) | 4.5 (2.4)
  Week 24 | 5.3 (2.0) | 4.6 (2.3) | 4.7 (2.7)

11. Secondary Outcome: General Health Visual Analog Scale (VAS)
Description: 100 mm line (VAS) marked by participant. Participants were asked, "How do you feel concerning your arthritis?" Total possible score range, 0 mm = very well to 100 mm = extremely bad.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 7
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks: 1) dress/groom; 2) arise; 3) eat; 4) walk; 5) reach; 6) grip; 7) hygiene; and 8) common activities over past week. Each item scored on 4-point Likert scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. The overall disability index computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
units on a scale
  Baseline | 1.8 (0.6) | 1.7 (0.6) | 1.6 (0.7)
  Week 2 | 1.5 (0.6) | 1.4 (0.7) | 1.3 (0.6)
  Week 4 | 1.4 (0.7) | 1.4 (0.7) | 1.3 (0.7)
  Week 8 | 1.5 (0.7) | 1.3 (0.6) | 1.2 (0.7)
  Week 12 | 1.5 (0.7) | 1.3 (0.6) | 1.1 (0.7)
  Week 16 | 1.4 (0.7) | 1.2 (0.6) | 1.1 (0.7)
  Week 20 | 1.4 (0.7) | 1.2 (0.7) | 1.0 (0.8)
  Week 24 | 1.4 (0.6) | 1.2 (0.7) | 1.0 (0.8)

13. Secondary Outcome: Disease Activity Score Based on 28-joints Count (DAS28)
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and participant's general health visual analog scale (scores ranging 0 [very well] to 100 mm [extremely bad]). DAS28 less than or equal to (=<) 3.2 = low disease activity, DAS28 greater than (>) 3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
units on a scale
  Baseline | 6.1 (0.7) | 5.8 (0.9) | 6.1 (1.0)
  Week 2 | 5.4 (1.0) | 5.1 (1.3) | 5.3 (1.3)
  Week 4 | 5.2 (1.1) | 4.9 (1.4) | 5.0 (1.4)
  Week 8 | 5.1 (1.3) | 4.6 (1.3) | 4.7 (1.3)
  Week 12 | 5.0 (1.3) | 4.3 (1.3) | 4.6 (1.4)
  Week 16 | 4.7 (1.5) | 3.9 (1.4) | 4.3 (1.4)
  Week 20 | 4.7 (1.4) | 4.0 (1.3) | 4.1 (1.4)
  Week 24 | 4.7 (1.4) | 4.1 (1.3) | 4.0 (1.5)

14. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Week 12, 24, 36, 52
Population: as for outcome 7
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns utility value for each domain in the profile. Score is transformed and results in total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 12, 24, 36, 52
Population: as for outcome 7
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Euro Quality of Life (EQ-5D)- Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Week 12, 24, 36, 52
Population: as for outcome 7
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Baseline, Week 12, 24, 36, 52
Population: as for outcome 7
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire: Rheumatoid Arthritis (WPAI-RA) Score
Description: WPAI-RA consisted of 6 items, a binary question on current employment, 3 questions on hours of work and work-loss, and 2 questions based on 0-10 point scale to judge how RA affects productivity at work and outside of work (0 = no effect on work and 10 = completely prevented from working). Four scores are derived: percent work time missed due to health, percent impairment while working due to health, percent overall work impairment due to health and percent activity impairment due to health. Total possible score range: 0 to 100, where 0 = no impairment and 100 = completely impaired.
Time Frame: Baseline, Week 12, 24, 36, 52
Population: as for outcome 7
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1.
Time Frame: Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TRU-015 Single Dose | TRU-015 Induction Dose
Number analyzed (Participants) | 74 | 75 | 73
percentage of participants
  Week 2: good response | 1.4 | 6.7 | 2.7
  Week 2: moderate response | 33.8 | 38.7 | 39.7
  Week 2: no response | 64.9 | 54.7 | 57.5
  Week 4: good response | 5.4 | 14.7 | 8.2
  Week 4: moderate response | 39.2 | 41.3 | 45.2
  Week 4: no response | 55.4 | 44.0 | 46.6
  Week 8: good response | 8.1 | 14.7 | 12.3
  Week 8: moderate response | 44.6 | 44.0 | 53.4
  Week 8: no response | 47.3 | 41.3 | 34.2
  Week 12: good response | 9.5 | 21.3 | 16.4
  Week 12: moderate response | 39.2 | 53.3 | 52.1
  Week 12: no response | 51.4 | 25.3 | 31.5
  Week 16: good response | 18.9 | 34.7 | 20.5
  Week 16: moderate response | 40.5 | 41.3 | 56.2
  Week 16: no response | 40.5 | 24.0 | 23.3
  Week 20: good response | 17.6 | 29.3 | 26.0
  Week 20: moderate response | 37.8 | 52.0 | 54.8
  Week 20: no response | 44.6 | 18.7 | 19.2
  Week 24: good response | 14.9 | 26.7 | 30.1
  Week 24: moderate response | 44.6 | 46.7 | 50.7
  Week 24: no response | 40.5 | 26.7 | 19.2
Statistical Analysis 1: Comparison: Placebo vs TRU-015 Single Dose; Week 2: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.106, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs TRU-015 Induction Dose; Week 2: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.322, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs TRU-015 Single Dose; Week 4 Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.059, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs TRU-015 Induction Dose; Week 4: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.250, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs TRU-015 Single Dose; Week 8: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.255, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs TRU-015 Induction Dose; Week 8: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.105, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs TRU-015 Single Dose; Week 12: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs TRU-015 Induction Dose; Week 12: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.019, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs TRU-015 Single Dose; Week 16: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.011, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Placebo vs TRU-015 Induction Dose; Week 16: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.113, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Placebo vs TRU-015 Single Dose; Week 20: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Placebo vs TRU-015 Induction Dose; Week 20: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Placebo vs TRU-015 Single Dose; Week 24: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Placebo vs TRU-015 Induction Dose; Week 24: Good response- A 2-sided CMH test, stratified by prior anti-TNF use and geographic region, was used; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Placebo (Part A): Placebo infusion, matched to TRU-015 (800 mg), IV along with methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at baseline. Placebo infusion, matched to TRU-015 (800 mg), IV along with methylprednisolone 100 mg or matching placebo IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of the infusion at Week 12. Participants in this group were assigned to either Placebo/TRU-SD or Placebo/TRU-ID in the Part B of the study.
- TRU-015 Single Dose (Part A): TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at baseline. Placebo infusion, matched to TRU-015 (800 mg), IV, methylprednisolone 100 mg or matching placebo IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of infusion at Week 12. Participants in this group were assigned to TRU-SD in the Part B of the study.
- TRU-015 Induction Dose (Part A): TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at baseline. TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule or matching placebo orally each day for 2 days prior to and on the morning of infusion at Week 12. Participants in this group were assigned to TRU-ID in the Part B of the study.
- TRU-015 Single Dose (Part B): TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 24. Placebo infusion, matched to TRU-015 (800 mg) IV along with placebo matched to methylprednisolone 100 mg IV 1 hr prior to infusion and placebo matched to prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 36.
- TRU-015 Induction Dose (Part B): Placebo infusion, matched to TRU-015 (800 mg), IV, placebo matched to methylprednisolone 100 mg IV 1 hr prior to infusion and placebo capsule matched to prednisone 20 mg orally each day for 2 days prior to and on the morning of infusion at Week 24. TRU-015 (800 mg) infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 36.
- Placebo/TRU-015 Single Dose (Part B): TRU-015 800 mg infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 24. Placebo infusion, matched to TRU-015 800 mg, IV, placebo matched to methylprednisolone 100 mg IV 1 hr prior to infusion and placebo capsule matched to prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 36.
- Placebo/TRU-015 Induction Dose (Part B): TRU-015 800 mg infusion IV, methylprednisolone 100 mg IV 1 hr prior to infusion and prednisone 20 mg capsule orally each day for 2 days prior to and on the morning of infusion at Week 24 and 36.
Arm/Group | Placebo (Part A) | TRU-015 Single Dose (Part A) | TRU-015 Induction Dose (Part A) | TRU-015 Single Dose (Part B) | TRU-015 Induction Dose (Part B) | Placebo/TRU-015 Single Dose (Part B) | Placebo/TRU-015 Induction Dose (Part B)
Serious Adverse Events (participants affected / at risk) | 7/74 | 4/75 | 7/73 | 2/56 | 2/55 | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 25/74 | 27/75 | 25/73 | 22/56 | 12/55 | 18/31 | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=74) | TRU-015 Single Dose (Part A) (N=75) | TRU-015 Induction Dose (Part A) (N=73) | TRU-015 Single Dose (Part B) (N=56) | TRU-015 Induction Dose (Part B) (N=55) | Placebo/TRU-015 Single Dose (Part B) (N=31) | Placebo/TRU-015 Induction Dose (Part B) (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=74) | TRU-015 Single Dose (Part A) (N=75) | TRU-015 Induction Dose (Part A) (N=73) | TRU-015 Single Dose (Part B) (N=56) | TRU-015 Induction Dose (Part B) (N=55) | Placebo/TRU-015 Single Dose (Part B) (N=31) | Placebo/TRU-015 Induction Dose (Part B) (N=32)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 4 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 4 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2
Bronchitis (Infections and infestations) | 4 | 2 | 0 | 1 | 1 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 4 | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 6 | 5 | 8 | 3 | 6 | 4
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 3 | 3 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 7 | 4 | 6 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 0 | 2 | 1 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7 | 5 | 1 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 10 | 3 | 2 | 3 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 5 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
As the results of the primary analysis did not meet the predefined efficacy criteria, the development of TRU-015 was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.